CLINICAL TRIAL: NCT03608384
Title: Characteristic of Drug Users Chronic Wound
Acronym: TOXIPO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS/TOXIPO-SCHMUTZ/ELR
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Wound; Drug Use
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to describe demographic, clinical, etiological characteristic and evolution of drug addict's chronic wounds .

ELIGIBILITY:
Inclusion Criteria:

* all drug addict with chronic wound ( evolving at least since 1 month)

Exclusion Criteria:

* use following medication inductor of cutaneous ulcer: hydroxycarbamide, gefitinib, cetuximab, sunitinib, sorafenib, pazopanib, gemcitabine, sirolimus, methotrexate, nicorandil .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Drug addict are mainly young man, use intravenous drug ( opioid, cocaine) and inhaled drug ( cannabis).
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
clinical venous insufficiency - presence of oedema | at inclusion
  presence of oedema

SECONDARY OUTCOMES:
clinical venous insufficiency - presence of varicose | at inclusion
  presence of varicose
clinical venous insufficiency - presence of white atrophy | at inclusion
  presence of white atrophy
clinical venous insufficiency - presence of varicose eczema | at inclusion
  presence of varicose eczema

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Schmutz, Study Director — CHRU Vandoeuvre-Lès-Nancy
Locations (1):
- CHRU De Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided